CLINICAL TRIAL: NCT03167463
Title: Stentless Endoscopic Transnasal Transseptal Choanoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Ezzat, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SETTC
Record Dates: First submitted 2017-05-18; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Otolaryngological Disease
MeSH Terms: conditions — Otorhinolaryngologic Diseases | interventions — Surgical Flaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- choanoplasty with flap (Experimental): flap surgery
  Interventions: Procedure: flap

INTERVENTIONS:
Procedure: flap — Repair choanal atresia with using flap during surgery

SUMMARY:
Congenital choanal atresia is an abnormality of the posterior nasal passages resulting in complete or partial obstruction of the nasal airways. It has an incidence of 1: 5000 to 8000 live births, with a female predominance. 41% - 72% occur in conjunction with non-syndromic facial abnormalities such as arched palate, cleft lip, and auricular deformities. About 4% present as a component of chromosomally-based syndromes such as (coloboma, heart defect, atresia choanae, retarded growth, genital abnormality, and ear abnormality" and Treacher Collins syndromes.

Previous reports have described the ratio of bony to membranous choanal atresia as 9:1. However, a detailed review of computed tomography study combined with histopathological studies has shown mixed bony-membranous atresia in about 70% of cases and purely bony atresia in 30% of cases.

DETAILED DESCRIPTION:
Common choanal atresia repair techniques include puncture and dilatation of the atretic area. Endoscopic drilling combined with dissection of the atretic plate and its surrounding structures has been introduced more recently. The approaches have been through transnasal, transpalatal, and transseptal routes. Each of which have experienced varying popularity through time. Regardless of the access route and repair technique used, re-stenosis is a common postoperative complication. To prevent re-stenosis and subsequent re-operation, many authors advocate meticulous preservation of mucosa for use as flaps, which in most cases are combined with postoperative stenting. However, stenting, is controversial

The surgical procedure is performed under general anesthesia. Preoperatively, cotton pledgets soaked in a solution of topical vasoconstrictors are placed against the nasal mucosa for topical decongestion. Local anesthesia is infiltrated into the nasal septum, the atretic plate, the middle turbinate, and the superolateral nasal wall. An endoscopic view of the surgical field is maintained at all times during the procedure using a 4-mm nasal endoscope with 0-degree or 30-degree visual angulation. Firstly, mucosa is elevated bilaterally from the underlying cartilaginous and bony septum on both sides. Then the posterior half of the septum including the vomer is removed using Blakesley forceps and a 1-mm or 2.5-mm diamond burr. After that, the flaps are fashioned using the preserved mucosa. At last, the flaps are secured in position with a thin layer of fibrin glue or gel foam. No packing or stenting is used. The patient is extubated immediately following the procedure and early oral feeding encouraged. The intended length of stay is overnight.

ELIGIBILITY:
Inclusion Criteria:

* • Denovo cases of unilateral congenital choanal atresia.

  * Revision cases of unilateral congenital choanal atresia.
  * Denovo cases of bilateral congenital choanal atresia.
  * Revision cases of bilateral congenital choanal atresia.

Exclusion Criteria:

* • Any associated medical comorbidity that contraindicates general anesthesia.

  * Refusal of enrollment in the research by care givers.

Ages: 3 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-19 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with postoperative relief of obstruction | 1 month
  number of patients will be cure after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Faculty of medicine Assiut University, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicin, Asyut, Assiut University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided